CLINICAL TRIAL: NCT05556512
Title: A Phase 3, Randomized, Double-blind, Placebo-Controlled Study to Investigate the Effect of Tirzepatide on the Reduction of Morbidity and Mortality in Adults With Obesity
Brief Title: A Study of Tirzepatide (LY3298176) on the Reduction on Morbidity and Mortality in Adults With Obesity
Acronym: SURMOUNT-MMO
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17253; I8F-MC-GPIJ (Other: Eli Lilly and Company); 2022-501744-15-00 (Other: EU Clinical Trial Number)
Record Dates: First submitted 2022-09-22; First posted 2022-09-27 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Obesity; Overweight
MeSH Terms: conditions — Obesity; Overweight | interventions — Tirzepatide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tirzepatide (Experimental): Participants will receive escalated doses of tirzepatide subcutaneously (SC) up to a maximum tolerated dose.
  Interventions: Drug: Tirzepatide
- Placebo (Placebo Comparator): Participants will receive tirzepatide matched placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tirzepatide — Administered SC
  Other Names: LY3298176
  Arms: Tirzepatide
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
This study will investigate the effect of tirzepatide on the reduction of morbidity and mortality in adults living with obesity and provide additional evidence for the potential clinical benefits of tirzepatide in this population.

ELIGIBILITY:
Inclusion Criteria:

* Have a body mass index (BMI) ≥27.0 kilogram/square meter (kg/m ²)
* Are either

  * individuals ≥40 years of age with established cardiovascular disease (CVD).

    * CVD is defined as meeting at least one of the following:

      * Coronary artery disease
      * Cerebrovascular disease
    * Peripheral arterial disease OR
    * individuals without established CVD but have the presence of cardiovascular (CV) risk factors (primary prevention)
    * women 55-69 years of age or men 50-64 years of age with at least 3 risk factors like tobacco use, dyslipidemia, hypertension at screening, or

      * women ≥70 years of age or men, ≥65 years of age with at least 2 risk factors at screening.

Exclusion Criteria:

* Have type 1 diabetes (T1D) or (T2D), history of ketoacidosis, or hyperosmolar state/coma
* Have laboratory evidence diagnostic of diabetes mellitus at screening of HbA1c ≥6.5% (≥48 millimole/mole (mmol/mol) or fasting glucose (FG) ≥126 milligram/deciliter (≥7.0 millimole/liter (mmol/L).
* Any one of the following CV conditions within 90 days prior to screening

  * MI
  * acute coronary syndrome
  * stroke
  * coronary or peripheral arterial revascularization procedure, which may also include carotid artery revascularization, or
  * acute decompensated heart failure
* Have a known clinically significant gastric emptying abnormality such as severe gastroparesis or gastric outlet obstruction or have undergone or currently planning any gastric bypass (metabolic) surgery or restrictive bariatric surgery. Note: Liposuction or abdominoplasty are not considered as gastric bypass procedures.
* Have a history of chronic or acute pancreatitis
* Have a family or personal history of medullary thyroid carcinoma or multiple endocrine neoplasia syndrome type 2.
* Have acute or chronic hepatitis, or clinical signs or symptoms of any other liver disease, or have elevated liver enzyme measurements, determined by the central laboratory at screening
* Have a presence or history of malignant neoplasms within the past 5 years prior to screening.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15374 (Actual)
Dates: Start 2022-10-11 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Time to First Occurrence of Any Component Event of Composite (All-Cause Death, Nonfatal Myocardial Infarction (MI), Nonfatal Stroke, Coronary Revascularization, or Heart Failure Events) | Up to 5 Years
  Time to first occurrence of any component event of composite, all-cause death, nonfatal MI, nonfatal stroke, coronary revascularization, or heart failure events that results in hospitalization or urgent visits.

SECONDARY OUTCOMES:
Time to Onset of Type 2 Diabetes (T2D) | Up to 5 Years
Change from Baseline in Estimated Glomerular Filtration Rate (eGFR) | Up to 5 Years
  In participants with high or very high risk chronic kidney disease
Time to First Occurrence of Any Component Event of Major Adverse Cardiovascular Events-3 (MACE-3) (CV Death, Nonfatal MI or Nonfatal Stroke) | Up to 5 Years
  Time to first occurrence of any component event of MACE-3 (CV death, nonfatal MI or nonfatal stroke)
Mean Change from Baseline Short Form-36 Version 2 (SF-36 v2) Acute Form Physical Functioning Domain Score | Baseline, 2 Years
  The SF-36 v2 acute, 1-week recall version is a 36-item generic, participant-administered measure designed to assess the following 8 domains (Physical Functioning, Role-Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role - Emotional, and Mental Health. Each domain is scored individually and further aggregated into 2 health component summary scores, physical component and mental component summary. Scoring of each domain and both summary scores are norm-based and presented in the form of T-scores, with a mean of 50 and standard deviation of 10; higher scores indicate better levels of function and/or better health.
Time to the Occurrence of All-cause Death | Up to 5 Years
Time to First Occurrence of CV Death | Up to 5 Years
Time to First Occurrence of MI | Up to 5 Years
Time to First Occurrence of Stroke | Up to 5 Years
Time to First Occurrence of Coronary Revascularization | Up to 5 Years
Time to First Occurrence Heart Failure (HF) Events | Up to 5 Years
  Time to first occurrence heart failure (HF) events that result in hospitalization or urgent visits
Time to First Occurrence of Hospitalization for Unstable Angina | Up to 5 Years
Time to first occurrence of Hospitalization or Urgent Visit | Up to 5 Years
  Time to first occurrence of hospitalization or urgent visit due to atrial fibrillation, or cardioversion or ablation for atrial fibrillation
Time to First Occurrence of Any Component Event of the Composite Endpoint (eGFR, ESRD, or Renal Death) | Up to 5 Years
  Time to first occurrence of any component event of the composite endpoint ≥40% sustained decline in eGFR, ESRD, or renal death.
Percent Change from Baseline in Body Weight | Baseline, 156 Weeks
Change from Baseline in Systolic Blood Pressure (SBP) in Millimeter Mercury (mmHg) | Baseline, 156 Weeks
Change from Baseline Diastolic Blood Pressure (DBP) (mmHg) | Baseline, 156 Weeks
Percentage of Participants with Hemoglobin A1c (HbA1c) <39 Millimole/Mole (mmol/mol) (5.7%) | Up to 5 Years
  Percentage of participants with HbA1c <39 mmol/mol (5.7%) at each time where HbA1c is assessed for participants with a screening HbA1c ≥39 mmol/mol.
Time to First Occurrence of Any Component Event of Composite Endpoint (All-Cause Death, Nonfatal MI, Nonfatal Stroke, Coronary Revascularization, Heart Failure Events, > 40% Sustained Decline in eGFR, or End Stage Renal Disease) | Up to 5 Years
  In participants with prediabetes

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559 or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (667):
- United States (164):
  - Prime Medical Group, LLC dba Gilbert Center for Family Medicine, LLC, Gilbert, Arizona
  - Aventiv Research, Mesa, Arizona
  - Elite Clinical Studies, Phoenix, Arizona
  - Pima Heart, Tucson, Arizona
  - KLR Business Group, Inc. dba Arkansas Clinical Research, Little Rock, Arkansas
  - Smart Cures Clinical Research, Anaheim, California
  - Kidney & Hypertension Center - Apple Valley, Apple Valley, California
  - Hope Clinical Research, Inc., Canoga Park, California
  - John Muir Physician Network Research Center, Concord, California
  - Neighborhood Healthcare Institute of Health, Escondido, California
  - HB Clinical Trials - Fountain Valley, Fountain Valley, California
  - Valiance Clinical Research, Huntington Park, California
  - Scripps Whittier Diabetes Institute, La Jolla, California
  - Velocity Clinical Research, San Diego, La Mesa, California
  - First Valley Medical Group, Lancaster, California
  - Long Beach Clinical Trials, Long Beach, California
  - Infinity Clinical Research - Norco, Norco, California
  - California Medical Research Associates, Northridge, California
  - Diabetes Associates Medical Group, Orange, California
  - University of California Irvine Medical Center, Orange, California
  - FOMAT Medical Research, Oxnard, California
  - Desert Oasis Healthcare Medical Group, Palm Springs, California
  - Dream Team Clinical Research, Pomona, California
  - Rancho Cucamonga Clinical Research, Rancho Cucamonga, California
  - Artemis Institute for Clinical Research, Riverside, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Acclaim Clinical Research, San Diego, California
  - Velocity Clinical Research, Santa Ana, Santa Ana, California
  - Valiance Clinical Research, Tarzana, California
  - Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center, Torrance, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Millennium Clinical Trials, Westlake Village, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Optum- Southwestern, Colorado Springs, Colorado
  - Kidney Associates of Colorado, Denver, Colorado
  - OptumCare Clinical Trials, LLC, Golden, Colorado
  - Clinical Research Consulting, Milford, Connecticut
  - Cardiology Associates of Fairfield County, P.C., Stamford, Connecticut
  - Chase Medical Research, LLC, Waterbury, Connecticut
  - Excel Medical Clinical Trials, Boca Raton, Florida
  - Encore Medical Research of Boynton Beach, Boynton Beach, Florida
  - Clinical Research of West Florida, Inc. (Clearwater), Clearwater, Florida
  - Northeast Research Institute (NERI), Fleming Island, Florida
  - Indago Research & Health Center, Inc, Hialeah, Florida
  - Northeast Research Institute - Downtown Office, Jacksonville, Florida
  - IHS Health Research, Kissimmee, Florida
  - Clinical Research of Central Florida, Lakeland, Florida
  - South Florida Clinical Research Institute, Margate, Florida
  - Felicidad Medical Research, Miami, Florida
  - Floridian Clinical Research, LLC, Miami Lakes, Florida
  - Florida Institute For Clinical Research, LLC, Orlando, Florida
  - Peace River Cardiovascular Center, Port Charlotte, Florida
  - Northeast Research Institute - St. Augustine, Saint Augustine, Florida
  - IMA Clinical Research St. Petersburg, St. Petersburg, Florida
  - Clinical Research of West Florida, Tampa, Florida
  - Metabolic Research Institute, Inc., West Palm Beach, Florida
  - Masters of Clinical Research, Augusta, Georgia
  - HOPE Clinical Research & Wellness, Conyers, Georgia
  - Center for Advanced Research & Education, Gainesville, Georgia
  - NSC Research, Johns Creek, Georgia
  - Balanced Life Health Care Solutions/SKYCRNG, Lawrenceville, Georgia
  - WR-Mount Vernon Clinical Research, LLC, Sandy Springs, Georgia
  - Rophe Adult and Pediatric Medicine/SKYCRNG, Union City, Georgia
  - North Georgia Clinical Research, Woodstock, Georgia
  - East-West Medical Research Institute, Honolulu, Hawaii
  - Elite Clinical Trials, Blackfoot, Idaho
  - Rocky Mountain Clinical Research, Idaho Falls, Idaho
  - Velocity Clinical Research, Boise, Meridian, Idaho
  - Solaris Clinical Research, Meridian, Idaho
  - IMA Clinical Research Chicago, Chicago, Illinois
  - Central Illinois Diabetes and Clinical Research a Division of Prairie Education and Research Cooperative, Springfield, Illinois
  - Healthcare Research Network - Chicago, Tinley Park, Illinois
  - American Health Network of Indiana, LLC - Avon, Avon, Indiana
  - Qualmedica Research, LLC, Evansville, Indiana
  - American Health Network of Indiana, LLC - Franklin, Franklin, Indiana
  - American Health Network of Indiana, LLC - Greenfield, Greenfield, Indiana
  - Iowa Diabetes and Endocrinology Research Center, West Des Moines, Iowa
  - Cotton O'Neil Diabetes & Endocrinology, Topeka, Kansas
  - Cotton O'Neil Mulvane, Topeka, Kansas
  - Qualmedica Research, Bowling Green, Kentucky
  - L-MARC Research Center, Louisville, Kentucky
  - Qualmedica Research, LLC, Owensboro, Kentucky
  - Ascension Saint Agnes Heart Care, Baltimore, Maryland
  - Centennial Medical Group, Columbia, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital Diabetes Program, Boston, Massachusetts
  - NECCR PrimaCare Research, Fall River, Massachusetts
  - ActivMed Practices and Research, Methuen, Massachusetts
  - Arcturus Healthcare , PLC, Troy Internal Medicine Research Division, Troy, Michigan
  - M Health Fairview St. John's Hospital, Maplewood, Minnesota
  - The National Diabetes & Obesity Research Institute, Diamondhead, Mississippi
  - Prime Health and Wellness/SKYCRNG, Fayette, Mississippi
  - Olive Branch Family Medical Center, Olive Branch, Mississippi
  - SKY Integrative Medical Center/SKYCRNG, Ridgeland, Mississippi
  - StudyMetrix Research, City of Saint Peters, Missouri
  - Healthcare Research Network - St. Louis, Hazelwood, Missouri
  - Clinvest Research LLC, Springfield, Missouri
  - IMA Clinical Research - St. Louis, St Louis, Missouri
  - Billings Clinic, Billings, Montana
  - VA Nebraska-Western Iowa Health Care System, Omaha, Nebraska
  - DaVita Clinical Research - Las Vegas, Las Vegas, Nevada
  - Excel Clinical Research, LLC, Las Vegas, Nevada
  - Palm Research Center Tenaya, Las Vegas, Nevada
  - Palm Research Center Sunset, Las Vegas, Nevada
  - Advanced Research Institute - Reno, Reno, Nevada
  - UniMed Center, East Brunswick, New Jersey
  - NJ MedCare & NJ Heart, Linden, New Jersey
  - Hassman Research Institute Marlton Site, Marlton, New Jersey
  - IMA Clinical Research Warren, Warren Township, New Jersey
  - IMA Clinical Research, Albuquerque, New Mexico
  - Albany Medical College, Division of Community Endocrinology, Albany, New York
  - Meridian Clinical Research, LLC, Binghamton, New York
  - NYU Langone Health, New York, New York
  - IMA Clinical Research, New York, New York
  - Rochester Clinical Research, LLC, Rochester, New York
  - Meridian Clinical Research, LLC, Vestal, New York
  - Lillestol Research, Fargo, North Dakota
  - Aventiv Research Inc, Columbus, Ohio
  - Alliance for Multispecialty Research, LLC, Norman, Oklahoma
  - The Corvallis Clinic, P.C., Corvallis, Oregon
  - Heritage Valley Medical Group, Inc., Beaver, Pennsylvania
  - Capital Area Research, LLC, Camp Hill, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Tristar Clinical Investigations, Philadelphia, Pennsylvania
  - Preferred Primary Care Physicians, Preferred Clinical Research-St. Clair, Pittsburgh, Pennsylvania
  - Cardiology Consultants of Philadelphia Yardley, Yardley, Pennsylvania
  - WR-Clinsearch, LLC, Chattanooga, Tennessee
  - Texas Diabetes & Endocrinology, P.A., Austin, Texas
  - Pinnacle Clinical Research, Austin, Texas
  - Dallas Diabetes Research Center, Dallas, Texas
  - Soma Clinical Trials, Denison, Texas
  - Medresearch Inc, El Paso, Texas
  - Diabetes and Thyroid Center of Ft. Worth, Fort Worth, Texas
  - Valley Institute of Research - Fort Worth, Fort Worth, Texas
  - AngioCardiac Care of Texas, PA, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Biopharma Informatic, LLC, Houston, Texas
  - Next Level Urgent Care, Houston, Texas
  - Research Physicians Network, LLC, Houston, Texas
  - Epic Clinical Research, Lewisville, Texas
  - Texas Institute for Kidney and Endocrine Disorders, Lufkin, Texas
  - Biopharma Informatic, LLC, McAllen, Texas
  - Texas Institute of Cardiology, PA, McKinney, Texas
  - Southern Endocrinology Associates, Mesquite, Texas
  - North Hills Family Medicine/North Hills Medical Research, North Richland Hills, Texas
  - Clinical Trials of Texas, LLC, San Antonio, Texas
  - Pinnacle Clinical Research, San Antonio, Texas
  - VIP Trials, San Antonio, Texas
  - Consano Clinical Research, LLC, Shavano Park, Texas
  - DaVita Clinical Research - North Houston, Shenandoah, Texas
  - Northwest Houston Heart Center, Tomball, Texas
  - Impact Research Institute, Waco, Texas
  - Texas Valley Clinical Research, Weslaco, Texas
  - Soma Clinical Trials, Wylie, Texas
  - Advanced Research Institute, Ogden, Utah
  - Advanced Research Institute - Sandy, Sandy City, Utah
  - Kalo Clinical Research, West Valley City, Utah
  - Dominion Medical Associates, Inc., Richmond, Virginia
  - National Clinical Research, Inc, Richmond, Virginia
  - Eastside Research Associates, Redmond, Washington
  - Rainier Clinical Research Center, Renton, Washington
  - Central Washington Health Services Association d/b/a Confluence Health, Wenatchee, Washington
  - IMA Clinical Research, Morgantown, West Virginia
  - St. Vincent Hospital d/b/a Prevea Health, Green Bay, Wisconsin
- Argentina (60):
  - CONEXA Investigacion Clinica S.A., Buenos Aires
  - Instituto Médico Especializado (IME), Buenos Aires
  - CEMEDIC, Buenos Aires
  - Centro Privado de Medicina Familiar / Mindout Research, Buenos Aires
  - Stat Research S.A., Buenos Aires
  - Investigaciones Medicas Imoba Srl, Buenos Aires
  - Centro de Investigaciones Metabólicas (CINME), Buenos Aires
  - Centro Médico Viamonte, Buenos Aires
  - Mautalen Salud e Investigación, Buenos Aires
  - Consultorio de Investigación Clínica EMO SRL, Buenos Aires
  - Asociación de Beneficencia Hospital Sirio Libanés, Buenos Aires
  - Centro Medico Dra. Laura Maffei- Investigacion Clinica Aplicada, Buenos Aires
  - Fundación Respirar, Buenos Aires
  - Glenny Corp. S.A., Buenos Aires
  - CENUDIAB, Buenos Aires
  - CEMEDIAB, C.a.b.a.
  - CEDIC, CABA
  - CIPREC, CABA
  - Centro Medico Privado CEMAIC, Capital
  - Hospital San Roque, Córdoba
  - Instituto de Investigaciones Clínicas Córdoba, Córdoba
  - Sanatorio Privado Duarte Quirós, Córdoba
  - Instituto Médico DAMIC, Córdoba
  - Centro Medico Privado San Vicente Diabetes, Córdoba
  - Clínica Privada Velez Sarsfield, Córdoba
  - CIDIM-Centro Integral de Diagnostico por Imagenes Marchegiani, Córdoba
  - Instituto Medico Strusberg, Córdoba
  - Centro de Investigaciones Clinicas Instituto del Corazon (CICIC), Córdoba
  - MICA - Medicina e Investigación Cardiometabólica, Del Viso
  - CIPADI - Centro Integral de Prevencion y Atencion en Diabetes, Godoy Cruz
  - Centro de Investigaciones Clínicas Baigorria, Granadero Baigorria
  - CIMeL Clinical Research, Lanús
  - Centro de Investigaciones Médicas Mar del Plata, Mar del Plata
  - Instituto de Investigaciones Clínicas Mar del Plata, Mar del Plata
  - Omega Salud, Mar del Plata
  - Instituto de Cardiología Wolff, Mendoza
  - CIAD Moron, Morón
  - DIM Clínica Privada, Ramos Mejía
  - Instituto Médico Río Cuarto, Río Cuarto
  - INECO Neurociencias Oroño, Rosario
  - Instituto de Investigaciones Clinicas Rosario, Rosario
  - Instituto Especialidades de la Salud Rosario, Rosario
  - Instituto Médico Catamarca IMEC, Rosario
  - Instituto Médico Fundación Grupo Colaborativo Rosario Investigación y Prevención Medica, Rosario
  - Laboratorio de Hemostasia y Trombosis, Rosario
  - Fundacion Estudios Clinicos, Rosario
  - Centro Polivalente de Asistencia e Investigacion Clinica - CER San Juan, San Juan
  - Centro de Investigaciones Médicas Tucuman, SAN M. de Tucuman
  - Centro Modelo de Cardiología, San Miguel de Tucumán
  - Clínica Mayo de Urgencias Médicas Cruz Blanca S.R.L, San Miguel de Tucumán
  - Investigaciones Clínicas Tucumán, San Miguel de Tucumán
  - Go Centro Medico San Nicolás, San Nicolás
  - Centro de Diagnóstico y Rehabilitación (CEDIR), Santa Fe
  - Centro de Investigaciones Clinicas del Litoral, Santa Fe
  - Centro de Salud e Investigaciones Médicas, Santa Rosa
  - Sanatorio Norte, Santiago del Estero
  - Centro de Investigaciones Medicas Temperley, Temperley
  - Sanatorio San Martin, Venado Tuerto
  - Clinica Central, Villa Regina
  - Instituto de Investigaciones Clinicas Zarate, Zárate
- Australia (21):
  - Nightingale Research, Adelaide
  - Royal Adelaide Hospital, Adelaide
  - Paratus Clinical Research Western Sydney, Blacktown
  - Box Hill Hospital, Box Hill
  - Royal Brisbane and Women's Hospital, Brisbane
  - Core Research Group, Brisbane
  - Paratus Clinical Research Canberra, Bruce
  - Emeritus Research, Camberwell
  - Victorian Heart Hospital, Clayton
  - Barwon Health, Geelong
  - Austin Health - Repatriation Hospital, Heidelberg West
  - Royal Hobart Hospital, Hobart
  - Advara HeartCare Joondalup, Joondalup
  - Paratus Clinical Research Central Coast, Kanwal
  - Logan Hospital, Meadowbrook
  - Baker IDI Heart and Diabetes Institute - Melbourne, Melbourne
  - The AIM Centre / Hunter Diabetes Centre, Merewether
  - GenesisCare - Murdoch - Murdoch Drive, Murdoch
  - Southern Adelaide Diabetes & Endocrine Services, Oaklands Park
  - University of Sydney - Charles Perkins Centre, Sydney
  - The Queen Elizabeth Hospital, Woodville
- Austria (7):
  - VIVIT, Feldkirch
  - Medizinische Universität Graz, Graz
  - Medizinische Universitaet Innsbruck, Innsbruck
  - Klinik Landstraße, Vienna
  - Zentrum für klinische Studien Dr Hanusch Gmbh, Vienna
  - Universitaetsklinikum Allgemeines Krankenhaus Wien, Vienna
  - Klinik Hietzing, Vienna
- Belgium (9):
  - AZORG Campus Aalst-Moorselbaan, Aalst
  - Imelda General Hospital, Bonheiden
  - Université Libre de Bruxelles - Hôpital Erasme, Brussels
  - Antwerp University Hospital, Edegem
  - UZ Gent, Ghent
  - Jessa Ziekenhuis, Hasselt
  - UZ Leuven, Leuven
  - Az Damiaan vzw, Ostend
  - AZ Nikolaas, Sint-Niklaas
- Brazil (28):
  - Centro de Pesquisa Clinica do Brasil, Brasília
  - Chronos Pesquisa Clínica, Brasília
  - Centro de Pesquisa Sao Lucas, Campinas
  - Instituto de Pesquisa clinica de Campinas, Campinas
  - Loema Instituto de Pesquisa Clinica, Campinas
  - Cline Research Center, Curitiba
  - Quanta Diagnóstico e Terapia, Curitiba
  - Centro de Diabetes Curitiba, Curitiba
  - Centro De Diabetes Metabolismo E Endocrinologia, Fortaleza
  - Centro de Pesquisas em Diabetes e Doenças Endócrino-Metabólicas, Fortaleza
  - Instituto Do Coracao De Marilia, Marília
  - CHN - Complexo Hospitalar de Niterói, Niterói
  - Núcleo de Pesquisa Clínica do Rio Grande do Sul, Porto Alegre
  - IBPClin - Instituto Brasil de Pesquisa Clínica, Rio de Janeiro
  - Pesquisare Saude, Santo André
  - Praxis Pesquisa Medica, Santo André
  - Centro Multidisciplinar de Estudos Clinicos, São Bernardo do Campo
  - ISPEM - Instituto São José dos Campos em Pesquisas Médicas, São José dos Campos
  - Instituto de Pesquisa Clinica, São Paulo
  - CPQuali Pesquisa Clínica, São Paulo
  - CPCLIN, São Paulo
  - NotreDame Intermedica Saude S.A, São Paulo
  - BR Trials - Ensaios Clinicos e Consultoria, São Paulo
  - Hospital 9 De Julho, São Paulo
  - CEPIC - Centro Paulista de Investigação Clínica, São Paulo
  - Hospital das Clinicas FMUSP, São Paulo
  - CEDOES, Vitória
  - Integral Pesquisa e Ensino, Votuporanga
- Canada (26):
  - LMC Clinical Research Inc. (Brampton), Brampton
  - C-health Research, Calgary
  - Ecogene-21, Chicoutimi
  - Med Trust Research, Courtice
  - Medicor Research, Greater Sudbury
  - Health Sciences North, Greater Sudbury
  - Viacar Recherche Clinique, Greenfield Park
  - NSHA-QEII Health Sciences Centre-Dickson Bldg, Halifax
  - Premier Clinical Trial Network, Hamilton
  - The Wharton Medical Clinic Clinical Trials Inc, Hamilton
  - Manna Research, Lévis
  - G A Research Associates, Moncton
  - Power Clinical Research, Montreal
  - Fraser Clinical Trials Inc, New Westminster
  - North York Diagnostic and Cardiac Centre, North York
  - Centricity Research Oshawa, Oshawa
  - Manna Research Montreal, Pointe-Claire
  - Alpha Recherche Clinique, Québec
  - ALPHA Recherche Clinique, Québec
  - Bluewater Clinical Research Group Inc., Sarnia
  - Synergy Medical Clinic, Sherwood Park
  - Centre de Medecine Metabolique de Lanaudiere (CMML), Terrebonne
  - LMC Clinical Research Inc. (Bayview), Toronto
  - Diabetes Heart Research Centre, Toronto
  - Dr. Anil K. Gupta Medicine Professional Corporation, Toronto
  - Dr. M.B. Jones Inc., Victoria
- China (32):
  - Peking University People's Hospital, Beijing
  - Beijing Friendship Hospital Affiliate of Capital University, Beijing
  - Beijing Pinggu District Hospital, Beijing
  - China-Japan Union Hospital, Changchun
  - Beijing Tsinghua Changgung Hospital, Changping
  - Chengdu Fifth People's Hospital, Chengdu
  - West China Hospital Sichuan University, Chengdu
  - Chongqing General Hospital, Chongqing
  - Hainan General Hospital, Haikou
  - The Fourth Affiliated Hospital of Harbin Medical University, Harbin
  - Hebei Medical University - Harrison International Peace Hospital, Hengshui Shi
  - First Huai'an Hospital Affiliated to Nanjing Medical University, Huai'an
  - Huzhou Central Hospital, Huzhou
  - Jinan Central Hospital, Jinan
  - The First People's Hospital of Yunnan Province, Kunming
  - Lanzhou university second hospital, Lanzhou
  - The First Affiliated Hospital of Henan University of Science &Technology, Luoyang Shi
  - The Third Hospital of Nanchang, Nanchang
  - Nanjing First Hospital, Nanjing
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing
  - Nanjing Medical University - Nanjing Jiangning Hospital, Nanjing
  - Third People's Hospital of Hainan Province, Sanya
  - Shanghai 9th People hospital, Shanghai
  - The People's Hospital of Liaoning Province, Shenyang
  - Siping Central People's Hospital, Siping
  - Tianjin Medical University General Hospital, Tianjin
  - Tianjin People' s Hospital, Tianjin
  - Wuhan University Medical College - Hubei Zhongshan Hospital, Wuhan
  - Wuxi People's Hospital, Wuxi
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - Shaanxi provincial people's hospital, Xi'an
  - The Second Affiliated Hospital of Zhengzhou University, Zhengzhou
- Czechia (14):
  - Kardiologicka ambulance, Brandýs nad Labem-Stará Boleslav
  - Nemocnice Cesky Krumlov, Český Krumlov
  - Asclepiades, Havířov
  - CTC Hodonin s.r.o., Hodonín
  - GAE s.r.o., Jindřichův Hradec
  - PreventaMed, Olomouc
  - Kardiologicka a Angiologicka Ambulance, Ostrava
  - Nefrologie, Prague
  - FaraCol s.r.o., Prague
  - Poliklinika Lípa Centrum, Prague
  - Kardiologicka ambulance s.r.o., Příbram
  - Angionika, Slaný
  - Kardiologicka ambulance MUDr. Ferkl s.r.o., Trutnov
  - Cardio Research, s.r.o, Zlín
- France (13):
  - Centre Hospitalier Sud Francilien, Corbeil-Essonnes
  - Chu Grenoble Alpes, La Tronche
  - Centre Hospitalier Louis Pasteur, Le Coudray
  - Hôtel-Dieu du Creusot - site Harfleur, Le Creusot
  - Centre Hospitalier Universitaire de Limoges - Hôpital Dupuytren, Limoges
  - Centre Hospitalier Universitaire de Nice - Hôpital l'Archet, Nice
  - Assistance Publique Hôpitaux de Paris - Groupe Hospitalier 10e - Hôpital Lariboisière, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Hôpital Nord Guillaume-et-René-Laennec / CHU de Nantes, Saint-Herblain
  - CHU Strasbourg-Hautepierre, Strasbourg
  - CHU Rangueil, Toulouse
  - Groupe Hospitalier Mutualiste Les Portes du Sud, Vénissieux
- Germany (21):
  - Kardiologische Praxis Dr. med. univ. Wolfgang Jungmair, Bad Homburg
  - Herz - und Diabeteszentrum Nordrhein - Westfalen, Bad Oeynhausen, Bad Oeynhausen
  - Klinische Forschung Berlin, Berlin
  - Universitaetsklinikum Carl Gustav Carus Dresden, Dresden
  - InnoDiab Forschung Gmbh, Essen
  - Medizentrum Essen Borbeck, Essen
  - Praxis am Markt - Dr. Bernd Becker, Essen
  - Universitätsklinikum Frankfurt Goethe-Universität, Frankfurt
  - ClinPhenomics CVC GmbH, Frankfurt
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau
  - Velocity Clinical Research Hamburg GmbH, Hamburg
  - Diabeteszentrum Hamburg West, Hamburg
  - AmBeNet GmbH, Leipzig
  - Diabetologikum Ludwigshafen/Die Praxis am Ludwigsplatz, Ludwigshafen am Rhein
  - Universität zu Lübeck - Institut für Endokrinologie und Diabetes, Lübeck
  - Institut für Diabetesforschung GmbH Münster, Münster
  - Arztpraxis Christine Kosch Pirna, Pirna
  - Zentrum für klinische Studien, Saint Ingbert
  - Universitaetsklinikum Tuebingen, Tübingen
  - Gemeinschaftspraxis Prof. Dr. med. Stephan Jacob, Dr. med. Frohmut Jacob, Villingen-Schwenningen
  - Praxis Sauter & Sauter & Vorbach, Wangen
- Greece (14):
  - General Hospital of Athens "G. Gennimatas", Athens
  - General Hospital of Athens Laiko, Athens
  - Athens Medical Center, Athens
  - Attikon General University Hospital, Chaïdári
  - University General Hospital of Heraklion, Heraklion
  - University Hospital of Ioannina, Ioannina
  - General Hospital of Lamia, Lamia
  - University General Hospital of Larissa, Larissa
  - Iatriko Paleou Falirou Medical Center, Palaió Fáliro
  - Thermi Clinic, Thermi,Thessaloniki
  - AHEPA University General Hospital of Thessaloniki, Thessaloniki
  - Euromedica General Clinic of Thessaloniki, Thessaloniki
  - Ippokrateio General Hospital of Thessaloniki, Thessaloniki
  - Papageorgiou General Hospital of Thessaloniki, Thessaloniki
- Hungary (18):
  - DRC Gyógyszervizsgáló Központ, Balatonfüred
  - Szent Margit Rendelintézet, Budapest
  - Clinexpert Kft., Budapest
  - Óbudai Egészségügyi Centrum, Budapest
  - Semmelweis University, Budapest
  - Dél-Pesti Centrumkórház, Budapest
  - Magyar Honvedseg Egeszsegugyi Kozpont, Budapest
  - TRANTOR'99 Bt. Anyagcsere Centrum, Budapest
  - Újpesti Egészségügyi Nonprofit Kft, Budapest
  - Strazsahegy Medicina Bt., Budapest
  - Bajcsy-Zsilinszky Kórház, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Kistarcsai Flor Ferenc Korhaz, Kistarcsa
  - Selye János Kórház, Komárom
  - Kanizsai Dorottya Korhaz, Nagykanizsa
  - Allergo-Derm Bakos Kft, Szolnok
  - Markusovszky Egyetemi Oktatokorhaz, Szombathely
  - Minoseg Orvoscsoport Kft, Veszprém
- India (10):
  - Gujarat Endocrin Pvt Ltd, Ahmedabad
  - Sardar Patel Medical College, Bikaner
  - Osmania General Hospital, Hyderabad
  - King George's Medical University, Lucknow
  - Dayanand Medical College and Hospital, Ludhiana
  - Sir JJ Group of Hospitals, Mumbai
  - Kingsway Hospitals (Best Multispeciality Hospital in Nagpur), Nagpur
  - G.B. Pant Institute of Postgraduate Medical Education & Research, New Delhi
  - Nirmal Hospital Pvt Ltd., Surat
  - Shri Bachubhai Dahyabhai Mehta Mahavir Heart Institute, Surat
- Israel (14):
  - Barzilai Medical Center, Ashkelon
  - Rambam Health Care Campus, Haifa
  - Linn Medical Center, Haifa
  - Edith Wolfson Medical Center, Holon
  - Hadassah Medical Center, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Galilee Medical Center, Nahariya
  - Rabin Medical Center, Petah Tikva
  - Rabin Medical Center - Hasharon Campus, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - Kaplan Medical Center, Rehovot
  - Clalit Health Services - Sakhnin Community Clinic, Sakhnin
  - Sourasky Medical Center, Tel Aviv
  - Yitzhak Shamir Medical Center, Ẕerifin
- Italy (14):
  - A.O.U.C. Policlinico di Bari, Bari
  - IRCCS - AOU di Bologna, Bologna
  - Azienda Ospedaliero Universitaria S.Anna, Ferrara
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - Ospedale Santa Maria Goretti, Latina
  - Azienda Ospedale - Università Padova, Padua
  - A.O.U. Policlinico Paolo Giaccone, Palermo
  - Azienda di Rilievo Nazionale e Alta Specializzazione Civico Di Cristina Benfratelli, Palermo
  - Azienda Ospedaliera Universitaria Pisana, Pisa
  - Fondazione Policlinico Universitario Campus Bio-Medico, Rome
  - Fondazione Policlinico Tor Vergata, Rome
  - IRCCS Policlinico San Donato, San Donato Milanese
  - Presidio Ospedaliero Ospedale Sant'Anna, San Fermo della Battaglia
  - Azienda Ospedaliero-Universitaria Città della Salute e della Scienza di Torino, Torino
- Japan (9):
  - Tokyo-Eki Center-building Clinic, Chūōku
  - Fukuoka Wajiro Hospital, Fukuoka
  - Rinku General Medical Center, Izumisano
  - Rakuwakai Otowa Hospital, Kyoto
  - Tokyo Saiseikai Central Hospital, Minatoku
  - Fukuoka Shinmizumaki Hospital, Onga-gun
  - AMC Nishiumeda Clinic, Osaka
  - Shimada Clinic - Osaka, Osaka
  - Uji-Tokushukai Medical Center, Uji
- Mexico (40):
  - Fundación Cardiovascular de Aguascalientes A.C., Aguascalientes
  - Investigacion En Salud Y Metabolismo Sc, Chihuahua City
  - Centro de Estudios de Investigacion Metabolicos y Cardiovasculares, Ciudad Madero
  - Centro de Investigación y Gastroenterología, Cuauhtémoc
  - Instituto de Diabetes, Obesidad y Nutricion, Cuernavaca
  - Medical Group Culiacan, Culiacán
  - Centro Para El Desarrollo de La Medicina Y de Asistencia Medica Especializada S.C., Culiacán
  - Lahoja. Asociacion Para La Investigacion Y La Farmacovigilancia, Durango
  - Instituto Jalisciense de Investigacion en Diabetes y Obesidad, Guadalajara
  - Diseno y Planeacion en Investigacion Medica, Guadalajara
  - Centro de Investigacion Medica Integral, Guadalajara
  - Universidad de Guadalajara, Guadalajara
  - Clinica de Investigacion en Reumatologia y Obesidad S. C., Guadalajara
  - CICEJ Centro de Investigación Clínica Endocrinológica de Jalisco S.C, Guadalajara
  - Private Practice - Dr. Arechavaleta Granell Maria del Rosario, Guadalajara
  - Private Practice - Dr. Francisco Gerardo Padilla, Guadalajara
  - Unidad de Investigación Clínica y Atención Médica HEPA, Guadalajara
  - Virgen Cardiovascular Research SC, Guadalajara
  - Investigación Médica Sonora, S.C., Hermosillo
  - Centro de Investigacion en Artritis y Osteoporosis SC, Mexicali
  - RM Pharma Specialists, Mexico City
  - Hospital de Jésus, I.A.P., Mexico City
  - Caimed Investigacion En Salud S.A. de C.V., Mexico City
  - Centro Especializado En Diabetes, Obesidad Y Prevencion De Enfermedades Cardiovasculares, Mexico City
  - Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran, Mexico City
  - EME RED Hospitalaria, Mérida
  - Medical Care and Research SA de CV, Mérida
  - Cardiolink Clin Trials, Monterrey
  - IMED Internal Medicine Clin Trials, Monterrey
  - Hospital Universitario "Dr. Jose Eleuterio Gonzalez", Monterrey
  - UBAM Unidad Biomedica Avanzada Monterrey, Monterrey
  - Eukarya PharmaSite, Monterrey
  - Centro de Estudios Clínicos de Querétaro (CECLIQ), Querétaro
  - PanAmerican Clinical Research - Querétaro - Avenida Antea, Querétaro
  - Unidad Médica para la Salud Integral, San Nicolás de los Garza
  - Centro de Investigacion Cardiovascular y Metabólica, Tijuana
  - Instituto Veracruzano en Investigación Clínica S.C., Veracruz
  - Arké SMO S.A de C.V, Veracruz
  - Consultorio de Medicina Especilizada del Sector Privado, Xalapa
  - Centro de Investigacion Medica de Occidente, S.C., Zapopan
- Netherlands (11):
  - Ziekenhuisgroep Twente, locatie Almelo, Almelo
  - Meander Medisch Centrum, Amersfoort
  - Reinier de Graaf Ziekenhuis, locatie Delft, Delft
  - Albert Schweitzer Ziekenhuis, locatie Dordwijk, Dordrecht
  - Treant, locatie Scheper Ziekenhuis, Emmen
  - General Practitioners Research Institute (GPRI), Groningen
  - Martini Ziekenhuis, Groningen
  - Spaarne Gasthuis, Haarlem Zuid, Haarlem
  - Elkerliek Ziekenhuis, Helmond
  - Franciscus Gasthuis & Vlietland, Locatie Gasthuis, Rotterdam
  - Ziekenhuis Rivierenland, Tiel
- Poland (23):
  - Osteo Medic sc A. Racewicz, J. Supronik, Bialystok
  - Legeartis - Poradnie Specjalistyczne, Bialystok
  - Niepubliczny Specjalistyczny Zaklad Opieki Zdrowotnej Osrodek Diabetologiczny Popula Spolka Cywilna, Bialystok
  - Centrum Medyczne NEUROMED, Bydgoszcz
  - NZOZ Centrum Medyczne KERmed, Bydgoszcz
  - INTERCOR, Bydgoszcz
  - Diab Serwis Popenda Spółka Jawna, Chorzów
  - Ambulatorium Sp. z o.o., Elblag
  - Centrum Kliniczno-Badawcze, Elblag
  - Centrum Badan Klinicznych PI-House sp. z o.o., Gdansk
  - Medyczne Centrum Diabetologiczno Endokrynologiczno Metaboliczne DIAB-ENDO-MET, Krakow
  - Centrum Terapii Wspolczesnej J. M. Jasnorzewska Spolka Komandytowo-Akcyjna, Lodz
  - CenterMed Lublin NZOZ, Lublin
  - Gabinety TERPA, Lublin
  - Ekamed, Lublin
  - Gaja Poradnie Lekarskie Maciej Wiza, Poznan
  - Nzoz Neuro-Kard Ilkowski i Partnerzy SPL, Poznan
  - Centrum Medyczne "Diabetika", Radom
  - NZOZ Przychodnia Specjalistyczna Andrzej Wittek, Henryk Rudzki, Ruda Śląska
  - NBR Polska, Warsaw
  - Centralny Szpital Kliniczny MSW w Warszawie, Warsaw
  - Wojewódzki Zespól Specjalistycznej Opieki Zdrowotnej, Wroclaw
  - 4 Wojskowy Szpital Kliniczny z Polikliniką SPZOZ, Wroclaw
- Puerto Rico (7):
  - Advanced Clinical Research, LLC, Bayamón
  - Dorado Medical Complex, Dorado
  - Puerto Rico Health Institute, Dorado
  - Manati Center for Clinical Research, Manatí
  - Puerto Rico Medical Research, Ponce
  - Research and Cardiovascular Corp., Ponce
  - GCM Medical Group, PSC - Hato Rey Site, San Juan
- Romania (25):
  - SC Minimed SRL, Bacau
  - CMI Cardiologie - Dr. Mercea Corina Delia, Baia Mare
  - CMI DNBM Dr. Pop Lavinia, Baia Mare
  - C.M.D.T.A. Neomed, Brasov
  - Nicodiab, Bucharest
  - Hightech Medical Services SRL-Centrul pentru Studiul Metabolismului, Bucharest
  - Centrul Medical NutriLife, Bucharest
  - Centrul Medical Endocrinologie si Diabet Dr. Paveliu, Bucharest
  - S.C. Cardiomed S.R.L., Craiova
  - Spitalul Clinic Județean de Urgență, Craiova
  - Milena Sante, Galați
  - Diamed Obesity, Galați
  - Centrul Medical Consultmed, Iași
  - Gama Diamed, Mangalia
  - Diabdana, Oradea
  - Centrul Medical Grandmed, Oradea
  - Sal Med Srl, Piteşti
  - Dianutrilife Medica, Ploieşti
  - Clinica Korall, Satu Mare
  - Policlinica Astra Sibiu, Sibiu
  - Centrul Medical Mediab, Târgu Mureş
  - Private Practice - Dr. Cristian Podoleanu, Târgu Mureş
  - Cabinet Medical Dr.Geru, Timișoara
  - Institutul de Boli Cardiovasculare Timișoara, Timișoara
  - Centrul Medical Medicalis, Timișoara
- Slovakia (7):
  - MediTask, Bratislava
  - JM-Interna s.r.o, Dolný Kubín
  - AMBORA s.r.o. Interna ambulancia, Martin
  - FUNKYSTUFF s.r.o., Nové Zámky
  - BENIMED s.r.o. Kardiologicka ambulancia, Piešťany
  - DIA-MED CENTRUM s.r.o., Púchov
  - PENTES s.r.o. Kardiologicka ambulancia, Žilina
- South Korea (8):
  - Korea University Ansan Hospital, Ansan-si
  - Pusan National University Hospital, Busan
  - Seoul National University Bundang Hospital, Seongnam
  - Kyung Hee University Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
  - Wonju Severance Christian Hospital, Wŏnju
- Spain (29):
  - CHUAC-Complejo Hospitalario Universitario A Coruña, A Coruña
  - Centro Periférico de Especialidades Bola Azul, Almería
  - Hospital Universitario de La Ribera, Alzira
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Osi Bilbao-Basurto, Bilbao
  - Complejo Hospitalario Universitario de Ferrol (CHUF)- Hospital Naval, Ferrol
  - Hospital Universitario San Cecilio, Granada
  - Complejo Asistencial Universitario de León - Hospital de León, León
  - Hospital Universitario Arnau de Vilanova de Lleida, Lleida
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Quirón Málaga, Málaga
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Central de Asturias, Oviedo
  - Clínica Juaneda, Palma de Mallorca
  - Clinica Universidad de Navarra, Pamplona
  - Hospital Universitario Quironsalud Madrid, Pozuelo de Alarcón
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna
  - Hospital Virgen del Camino, Sanlúcar de Barrameda
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Clínica nuevas Tecnologías en Diabetes y Endocrinología (NTDE), Seville
  - Hospital Quiron Infanta Luisa, Seville
  - Vithas Hospital Sevilla, Seville
  - Hospital Clinico de Valencia, Valencia
  - Hospital General Universitario de Valencia, Valencia
  - Hospital Universitario Doctor Peset, Valencia
  - Hospital Virgen de las Montañas, Villamartín
- Taiwan (11):
  - Hsinchu Mackay Memorial Hospital, Hsinchu
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Chang Gung Memorial Hospital at Kaohsiung, Kaohsiung Niao Sung Dist
  - Far Eastern Memorial Hospital, New Taipei City
  - Taipei Medical University Shuang Ho Hospital, New Taipei City
  - Mackay Memorial Hospital -Tamshui Branch, New Taipei City
  - National Cheng Kung University Hospital, Tainan
  - Chi Mei Medical Center, Tainan
  - Taipei Medical University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
- Turkey (Türkiye) (17):
  - Çukurova Üniversitesi Tıp Fakültesi Adana Hastanesi, Adana
  - Ankara Universitesi Tip Fakultesi Hastanesi, Ankara
  - Akdeniz Universitesi Hastanesi, Antalya
  - Adnan Menderes University Medical Faculty, Aydin
  - Dokuz Eylül Üniversitesi, Balçova
  - Ege Universitesi Hastanesi, Bornova
  - Pamukkale University Medical Faculty, Fahri Goksin Oncology Centre, Denizli
  - Gaziantep Universitesi Sahinbey Arastirma ve Uygulama Hastanesi, Gaziantep
  - TC Saglik Bakanligi Goztepe Prof. Dr. Suleyman Yalcin Sehir Hastanesi, Kadıköy
  - Erciyes University Medical Faculty, Kayseri
  - Necmettin Erbakan Meram Medical Fac., Konya
  - Inonu Universitesi Turgut Ozal Tıp Merkezi, Malatya
  - Mersin University, Mersin
  - Sisli Etfal Training and Research Hospital, Sarıyer
  - Cumhuriyet Universitesi, Sivas
  - Baskent University Dr. Turgut Noyan Research and Training Center, Yüreğir
  - Bursa Yüksek İhtisas Eğitim Ve Araştırma Hastanesi, Yıldırım
- United Kingdom (15):
  - Oakenhurst Medical Practice, Blackburn
  - Southmead Hospital, Bristol
  - University Hospital Coventry & Warwickshire, Coventry
  - Ninewells Hospital and Medical School, Dundee
  - Staploe Medical Centre, Ely
  - Fowey River Practice, Fowey
  - Hull Royal Infirmary, Hull
  - Ipswich Hospital, Ipswich
  - Leicester General Hospital, Leicester
  - Royal Victoria Infirmary, Newcastle upon Tyne
  - Knowle House Surgery, Plymouth
  - Wickersley Health Centre - Clifton Medical Centre, Rotherham
  - Lister Hospital, Stevenage
  - Rame Group Practice, Torpoint
  - The Royal Cornwall Hospital, Truro

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- See also: A Study of Tirzepatide (LY3298176) on the Reduction on Morbidity and Mortality in Adults With Obesity (SURMOUNT-MMO) — https://trials.lilly.com/en-US/trial/362220